CLINICAL TRIAL: NCT06475482
Title: Development of a Novel Polyherbal Lip Hydrant for Improving Biophysical Barrier of the Lips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREC-DCU2023-060
Record Dates: First submitted 2024-02-15; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-02

CONDITIONS: Cheilitis
Keywords: Cheilitis; Aging; Lip roughness; Prevention
MeSH Terms: conditions — Cheilitis

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, controlled trial will be conducted at the Faculty of Dentistry, Chulalongkorn University. The 66 participants will be randomly assigned to receive either lip hydrant containing peppermint oil, perilla frutescens, and Emblica fruit extract or petroleum gel. Both lip products will be given to allocated participants in the product container of identical appearance. Both subjects and investigators will be blinded to the study randomization.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Petroleum gel (Vaseline) (Placebo Comparator): control group
  Interventions: Other: Petroleum gel
- Lip hydrant (Active Comparator): experimental group
  Interventions: Other: Lip hydrant

INTERVENTIONS:
Other: Lip hydrant — lip hydrant containing peppermint oil, perilla frutescens, and Emblica fruit extract or petroleum gel.
  Arms: Lip hydrant
Other: Petroleum gel — Vaseline
  Arms: Petroleum gel (Vaseline)

SUMMARY:
* The goal of this clinical trial is to evaluate the efficacy of the novel polyherbal lip hydrant on dryness, fine lines and color of the lips in 66Thai people aged between 18-40 years old. The inclusion criteria will include subjects with subjective complaint of dry lips.The main question it aims to answer is Does the novel polyherbal lip hydrant improve biophysical barrier of the lips?
* Participant will be asked to apply the lip hydrant or the petroleum gel once a day before bedtime, and refrain from using other lip products throughout the clinical trial period (28 days).
* Researchers will compare control group (Petroleum gel) with lip hydrant group to see whether biophysical barrier (wrinkles, colors, fine lines, roughness) improve or not.

ELIGIBILITY:
Inclusion Criteria:

* subjects with subjective complaint of dry lips;
* agree to comply with the study protocol
* agree not to apply any other products such as lipstick, lip gloss, lip conditioner to the lips other than the test product for the duration of the study
* provide a written informed consent prior to study enrollment.

Exclusion Criteria:

* Participants those having visible skin conditions which might interfere with the outcome assessment
* having a history of sensitivities to cosmetics products, or moisturizers; - having a known or suspected intolerance or hypersensitivity to herbal products or any of its ingredient
* taking medication or under the care of a doctor for one month prior to the commencement of the study, and throughout the entire test period
* having other types of cheilitis except cheilitis simplex.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Objective evaluation | 30 minutes per 1 participant
  Objective evaluation; using
  * Fotofinder to take a photograph of the lips.
  * Modified visual assessment scale to assess lip roughness score divided to 4 levels (1=not dry 2= dry without desquamated 3 = dry with slightly desquamated 4 = dry with heavy desquamated) and lip wrinkle score divided into 3 levels (1 = Almost no vertical wrinkle 2 = No deep vertical wrinkle 3= Many deep vertical wrinkle)
  * Antera 3D. (Texture, wrinkle, melanin pigment and hemoglobin) the value from Antera appear as the number with no unit,
  * Digital camera to evaluate overall clinical improvement of the lips

SECONDARY OUTCOMES:
Subjective evaluation | 5 minutes per 1 participant
  will be assessed at day 0 (baseline), day 1 and day 28 by using a self-reported questionnaire in scale from 1-10 points for patient's dry lip score which higher score means more dry lip feeling

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamura E, Ishikawa J, Yasuda Y, Yamamoto T. The efficacy of synthetic pseudo-ceramide for dry and rough lips. Int J Cosmet Sci. 2021 Apr;43(2):158-164. doi: 10.1111/ics.12677. Epub 2021 Mar 31. PMID 33258166
- [Background] Tamura E, Yasumori H, Yamamoto T. The efficacy of a highly occlusive formulation for dry lips. Int J Cosmet Sci. 2020 Feb;42(1):46-52. doi: 10.1111/ics.12583. PMID 31571236
- [Background] Trookman NS, Rizer RL, Ford R, Mehta R, Gotz V. Clinical assessment of a combination lip treatment to restore moisturization and fullness. J Clin Aesthet Dermatol. 2009 Dec;2(12):44-8. PMID 20725584
- [Derived] Sutthiboonyapan P, Sriratanasak N, Innets B, Angkanaporn N, Suntornchot P, Panyain W, Porntaveetus T, Wiriyakijja P, Chanvorachote P. A Randomized Double-Blind Controlled Evaluation of the Therapeutic Benefits of an Herbal Lip Hydrant. J Cosmet Dermatol. 2025 Mar;24(3):e70041. doi: 10.1111/jocd.70041. PMID 40013415